CLINICAL TRIAL: NCT00911196
Title: Analysis of the Incidence of Expression of Tumor Antigens and Tumor Marker in Cancer Tissue From Asian Patients With Hepatocellular Carcinoma and Evaluation of Prognostic Significance of These Tumor Antigens.
Brief Title: Analysis of Expression of Specific Markers and Their Prognostic Significance in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111726
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Prognosis; Markers; Expression analysis; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — This retrospective study is based upon the analysis of archived samples and patient-related data already available at the investigational site

GROUPS / COHORTS (1):
- Group A
  Interventions: Other: Retrospective analysis of already archived samples

INTERVENTIONS:
Other: Retrospective analysis of already archived samples — Analysis using RNA extracted from tissue samples already archived; Analysis by Fluorescent in situ hybridization (FISH) using tissue samples already archived.

SUMMARY:
Hepatocellular carcinoma is an aggressive disease with limited therapeutic options. Therefore, new approaches to treat this type of cancer are needed with immunotherapy potentially being one of these. As a first step in the development of novel therapies, expression analysis of specific markers, including tumor antigens will be carried out, and the correlation of expression with disease variables and clinical outcome will be assessed. This will be done retrospectively using archived hepatocellular carcinoma tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* The patient has pathologically proven hepatocellular carcinoma (any stage)
* All the data required are available from patient's records

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The proportion of hepatocellular carcinoma patients whose tumor tissue expresses specific tumor antigens. | At the time of analysis
The prognostic character of the expression of the tumor antigens | At the time of analysis
Expression of c-MET in the same hepatocellular carcinoma tumor samples | At the time of analysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Taipei, Taiwan
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai